CLINICAL TRIAL: NCT04980794
Title: Effectiveness of an Empirically Supported Family Intervention: Mental Health Outcomes, Mechanisms of Effect, and Organizational Factors
Brief Title: The Happy Families Project: Testing the Effectiveness of a Conflict Resolution Program for Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-0852
Record Dates: First submitted 2021-07-13; First posted 2021-07-28 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Mental Health; Conflict
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two conditions.
Who Masked: Participant
Masking Description: Participants are blind to condition assignments during their involvement in the program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parent-Child Intervention (Experimental): This is a four-dose intervention that includes psychoeducational modules and communication coaching administered through community organizations over the course of four weeks. Both participating adults and the participating child receive materials to review each week, paired with weekly contact from a family coach.
  Interventions: Behavioral: Parent-child intervention
- Self-study intervention (Active Comparator): This is a four-dose intervention that include written self-study materials to review, paired with weekly contact with a family coach. Both participating adults receive self-study materials; the participating child does not receive separate materials.
  Interventions: Behavioral: Self-study Intervention

INTERVENTIONS:
Behavioral: Parent-child intervention — Families (two adult caregivers, child between 4 and 17) receive four interactive, asynchronous psychoeducation modules to review on their own paired with weekly contact with a communication coach and two live sessions with a communication coach to discuss psychoeducation, receive feedback on their interactions, and practice a communication technique.
  Arms: Parent-Child Intervention
Behavioral: Self-study Intervention — Families (two adult caregivers) receive information in a newsletter format to review on their own, paired with weekly contact from a communication coach to answer questions and direct their attention toward specific topics in the newsletter.
  Arms: Self-study intervention

SUMMARY:
This study is designed to test the effectiveness of a psychoeducation-based program to address communication and conflict resolution in families, thereby supporting mental health in children and their caregivers.

DETAILED DESCRIPTION:
The goal of the study is to evaluate the effectiveness of a program to improve mental health in families by reducing stress and supporting effective communication and conflict resolution.

Families will be randomly assigned to one of two conditions: in the self-study condition, families will receive information to review on their own, paired with regular (weekly) contact from a family coach; in the second condition, families will receive information to review on their own, regular contact from a coach, and will participate in video sessions with a family coach who will provide feedback on their interactions and coaching on their use of a communication technique. Data collection, management and analysis will be conducted by researchers at the University of Notre Dame, but the intervention will occur through community organizations in three cities in Indiana, allowing for tests of the effectiveness of the program when it is implemented in community settings. Families will participate in a pre-test assessment, a four-week intervention, a post-test assessment, and a one-year follow up assessment. Also evaluated will be organizational factors and factors that impact ultimate implementation and scalability of the program in community settings.

ELIGIBILITY:
Inclusion Criteria:

* Two parents or primary caregivers
* Child between 4 and 17 years old
* English literate
* Able/willing to participate through the 12-month follow up assessment.

Exclusion Criteria:

* Families who cannot communicate in English
* Single parent families

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | 1 year
  Youth Adjustment
Center for Epidemiological Studies Depression Scale (CESD) | 1 year
  Youth Adjustment
Revised Children's Manifest Anxiety Scale (RCMAS) | 1 year
  Youth Adjustment
Child Behavior Checklist (CBCL) | 1 year
  Youth Adjustment
O'Leary Porter Scale (OPS) | 1 year
  Interadult Conflict
Family Interactions Coding Scale | 1 year
  Observational measures of interadult and family conflict
Security in the Marital System Questionnaire (SIMS-PR) | 1 year
  Youth Emotional Security: Testing process models associated with youth emotional security as the mechanism of effect for program effectiveness
Security in the Subsystem (SIS) | 1 year
  Youth Emotional Security: Testing process models associated with youth emotional security as the mechanism of effect for program effectiveness
Security in the Family System (SIFS) | 1 year
  Youth Emotional Security: Testing process models associated with youth emotional security as the mechanism of effect for program effectiveness
Organizational Characteristics Measure (purpose created measure of organizational characteristics) | 4 years
  Testing organizational factors associated with program effectiveness
Leadership Perspective Measure (purpose created measure of organizational leaderships' perspective on program, implementation and sustainability) | 4 years
  Testing organizational factors associated with program effectiveness
Facilitator Perspective Measure (purpose created measure of community facilitators' perspective on program implementation and training) | 4 years
  Testing organizational factors associated with program effectiveness

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Fort Wayne Center for Children and Families, Fort Wayne, Indiana
  - Indianapolis Virtual Site, Indianapolis, Indiana
  - University of Notre Dame, Notre Dame, Indiana

IPD SHARING:
Plan to Share IPD: Undecided